CLINICAL TRIAL: NCT01717781
Title: Prospective Randomized Trial on Laparoscopic Radical Hysterectomy With Pelvic Lymphadenectomy for the Treatment of Early Stage Cervical Cancer (FIGO Stages IA2-IB1-IIA<2cm) and Advanced Stage Cervical Cancer (FIGO Stages IB2-IIA>2 Cm-IIB) Submitted to NACT With Complete Clinical Response: Thunderbeat Technology Versus Standard Bipolar Electro Surgery
Brief Title: Thunderbeat Technology vs Standard Bipolar Electro Surgery in Laparoscopic Radical Hysterectomy and Pelvic Lymphadenectomy for Cervical Cancer
Acronym: Thunder Cervix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Director, Dip per la Tutela della Salute della Donna e della Vita Nascente, del Bambino e dell'Adolescente - Policlinico Gemelli, Rome, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Thunder Cervix
Record Dates: First submitted 2012-10-28; First posted 2012-10-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Cervical Cancer
Keywords: operative time; laparoscopy; radical hysterectomy; pelvic lymphadenectomy; cervical cancer; thunderbeat
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thunderbeat (Experimental): Laparoscopic radical hysterectomy with pelvic lymphadenectomy are performed with Thunderbeat technology: using Thunderbeat technique, surgeons can avoid changing instruments during surgery since Thunderbeat combines bipolar energy for haemostasis and ultrasound for dissection and cut.
  Thunderbeat is used to divide the round ligaments, to seal ovarian pedicles, to open the anterior and posteriors leaves of the broad ligaments peritoneum, to incise the bladder peritoneum, to develop the paravesical and pararectal spaces, to seal uterine arteries and uterine pedicles, to dissect the bladder and develop rectovaginal septum, to unroof the ureter, to cut parametria, and to divide the uterosacral ligaments. Monopolar hook is used in the culdotomy. Thunderbeat is also used to perform pelvic lymphadenectomy.
  Interventions: Procedure: Thunderbeat technology
- Standard (Active Comparator): Laparoscopic radical hysterectomy with pelvic lymphadenectomy are performed with standard bipolar electrosurgery.
  A 10 mm port is inserted at the umbilicus for the telescope. Once pneumoperitoneum (12 mmHg) is achieved, intra-abdominal visualization will be obtained with a 0° high-definition telescope.
  Two additional 5 mm ports are placed under direct visualization. One more 5-mm trocar is inserted in the right mid abdomen at the level of the umbilicus. The instruments used include bipolar grasper, monopolar scissors, monopolar hook, various graspers and a suction irrigation system.
  Interventions: Procedure: Standard bipolar electrosurgery

INTERVENTIONS:
Procedure: Thunderbeat technology
  Arms: Thunderbeat
Procedure: Standard bipolar electrosurgery
  Arms: Standard

SUMMARY:
This prospective randomized pilot study is aimed to verify if the operative time of a LRH with pelvic lymphadenectomy for early stage cervical cancer (FIGO stages IA2-IB1-IIA<2cm) and for advanced stage cervical cancer (FIGO stages IB2-IIA>2cm-IIB) submitted to neoadjuvant chemotherapy with complete clinical response could be reduced using Thunderbeat (an ultrasonic energy device that incises and coagulates by using ultrasonic and bipolar technology ) (Olympus Medical Systems Corp, Tokyo) vs. bipolar electrosurgery .

Secondary endpoints of this comparison are incidence of intra- or postoperative complications, estimated blood loss, postoperative pain, days of hospitalization and costs for the health care system.

DETAILED DESCRIPTION:
Radical abdominal hysterectomy (RAH) with pelvic lymphadenectomy is the standard surgical treatment for early stage cervical carcinoma FIGO stages IA2-IB1-IIA<2cm1. Since the early 90's laparoscopic radical hysterectomy with pelvic lymphadenectomy (LRH) has been suggested as surgical approach for the treatment of cervical cancer. In the recent years, many institutions have begun to consider it an attractive technique and to study its feasibility and safety. Most of these studies have shown that LRH is relatively more time-consuming than standard laparotomy and ranges from 90 to 420 minutes according to surgeons' experience and different techniques adopted to achieve hemostasis, resect the parametrium and uterosacrals. Spirtos et al. demonstrated that staplers could reduce mean operation time from 253 to 205 minutes if compared to argon beam coagulator. Moreover, the pulsed bipolar system was associated with significant reduction in operative time in comparison with the conventional bipolar system (mean, 172 minutes vs 229 minutes; P < 0.001). The largest series of LRH reported from a single institution by Puntambekar et al included 248 patients and described the "Pune technique" (anterior and posterior peritoneal U cuts, early dissection of the rectovaginal space, fully mobilization of the uterus, resection of the cardinal and uterosacral ligaments with Ligasure system (Ligasure Vessel Sealing System; Valleylab, Tyco Healthcare, Boulder, CO)), obtaining a very short mean operative time (mean, 92 minutes; range 6-120 minutes).

A recent review on laparoscopic and robot-assisted radical hysterectomy with pelvic lymphadenectomy including 17 studies reported a mean operating time of 202 minutes [range, 184-221 minutes] in the group of LRH, which matches with our experience of 210 min (range 180-240), using conventional bipolar electrosurgery.

The aim of this pilot RCT is to verify if the operative time of a LRH with pelvic lymphadenectomy for early stage cervical cancer (FIGO stages IA2-IB1-IIA<2cm) and for advanced stage cervical cancer (FIGO stages IB2-IIA>2cm-IIB) submitted to neoadjuvant chemotherapy (NACT) with complete clinical response could be further reduced using Thunderbeat (an ultrasonic energy device that incises and coagulates by using ultrasonic and bipolar technology ) (Olympus Medical Systems Corp, Tokyo) vs. bipolar electrosurgery .

Saving operative time would mean shorter anesthesia and faster recovery, further improving the safety profile of the laparoscopic approach in the treatment of cervical cancer.

Secondary endpoints of this comparison are incidence of intra- or postoperative complications (Cardiac, Respiratory, Neurological, Gastrointestinal, Renal, Fever, Wound or other Infection, Lymphocele), estimated blood loss, postoperative pain (evaluated by VAS), days of hospitalization and costs for the health care system.

ELIGIBILITY:
Inclusion/exclusion criteria

* Age ≤ 75 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* No actual pregnancies or P.I.D.
* No previous major abdominal surgical procedures For diseases
* Early stage cervical cancer (FIGO stages IA2-IB1-IIA<2cm) and advanced stage cervical cancer (FIGO stages IB2-IIA>2cm-IIB) submitted to NACT with complete clinical response
* No previous radiotherapy on the pelvic field
* No uterine size larger than conform 10 weeks gestation

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Operative time for laparoscopic radical hysterectomy with pelvic lymphadenectomy | 24 months
  Operative time will be calculated from the entrance in the abdominal cavity to the closure of the skin trocar accesses.

SECONDARY OUTCOMES:
Intra- or post operative complications | 24 months
  Cardiac, Respiratory, Neurological, Gastrointestinal, Renal, Fever, Wound or other Infection, Lymphocele

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred the Hearth, Rome, Italy, Italy